CLINICAL TRIAL: NCT00356486
Title: Open, Multicentre and Randomised Phase IV Study to Evaluate Viral Kinetics in the First 12 Weeks of Patients With Chronic Hepatitis C Genotypes 1 and 4 Coinfected by the Human Immunodeficiency Virus Treated With Induction Doses of Peginterferon Alpha-2a (40 KD) (270 μg/Week) and Ribavirin (1600 mg/Day) With Epoetin β Support (450 IU/kg/Week)
Brief Title: Viral Kinetics of Treatment With Peginterferon Alpha-2a, Ribavirin and Epoetin β in Patients Coinfected HCV/HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORAL-2; 2004 - 000907 -16
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Chronic Hepatitis C; Co-infection; Induction dose; HIV; HIV Infections
MeSH Terms: conditions — HIV Infections; Hepatitis C, Chronic; Coinfection | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Peginterferon alfa-2a (40 KD) (270 µg/week) + Ribavirin (1600 mg/day) + epoetin-β (450 UI/kg/week) for 4 weeks. Peginterferon alfa-2a (40 KD) (180 µg/week) + Ribavirin (1000-1200 mg/day) for 8 weeks
  Interventions: Drug: Peginterferon alfa-2a, Ribavirin, epoetin-β
- B (Experimental): Peginterferon alfa-2a (40 KD) (180 µg/week) subcutaneous + Ribavirin(1000-1200 mg/day) oral/day for 12 weeks
  Interventions: Drug: Peginterferon alfa-2a + Ribavirin for 12 weeks

INTERVENTIONS:
Drug: Peginterferon alfa-2a, Ribavirin, epoetin-β — Peginterferon alfa-2a(270 µg/week) + Ribavirin (1600 mg/day) + epoetin-β (450 UI/kg/week) for 4 weeks. Peginterferon alfa-2a (180 µg/week) + Ribavirin(1000-1200 mg/day) for 8 weeks
  Arms: A
Drug: Peginterferon alfa-2a + Ribavirin for 12 weeks — Peginterferon alfa-2a (40 KD) (180 µg/week) subcutaneous + Ribavirin(1000-1200 mg/day) oral/day for 12 weeks
  Arms: B

SUMMARY:
The purpose of this study is to compare the early virological response (EVR = undetectable [ribonucleic acid-hepatitis C virus] RNA-HCV or a reduction of > 2 log10) of patients with chronic hepatitis C coinfected with HIV treated with induction doses of peginterferon alpha-2a (40 KD) 270 µg/week and ribavirin 1600 mg/day for 4 weeks, followed by 8 weeks of treatment with peginterferon alpha-2a (40 KD) 180 µg/week and ribavirin 1000-1200 mg/day versus treatment with peginterferon alpha-2a (40 KD) 180 µg/week and ribavirin 1000-1200 mg/day for 12 weeks.

DETAILED DESCRIPTION:
This study seeks to ascertain whether treatment with higher doses of PEGASYS (270 µg/week) and ribavirin (1600 mg/day) for the first four weeks achieves the plasma concentrations of the product in the blood needed to reduce the half-life of the virions and accelerate the elimination thereof. This would bring the viral kinetic curves in coinfected patients closer to the model described for mono-infected HCV patients, probably achieving improved rates of response in week 12 (early virological response) and posterior in week 72 (sustained virological response).

Therefore, the patients were randomised to treatment with two different doses, 270 µg and 180 µg of PEGASYS, and 1600 mg and 1000-1200 mg of ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Serological evidence of chronic hepatitis C infection in an anti-HCV antibody test
* Detectable RNA-HCV plasma level genotype 1 and 4
* ALT serum activity above the upper limit of normality
* Chronic liver disease consistent with chronic hepatitis C infection in a biopsy obtained during the two years prior to inclusion in the study
* Serological evidence of HIV-1 infection, diagnosed by Enzyme-Linked Immunosorbent Assay (ELISA) and confirmed by Western-blot.
* Patients with CD4 cell count > 200 /µl
* Stable status in HIV-1 infection, in the investigator's opinion, in other words, patients that are not expected to progress during the study.
* Patients treated with stable anti-retroviral therapy (HAART), which does not include nucleoside analogues, for at least 6 weeks before the baseline assessment
* Patients that do not receive HAART therapy
* Negative pregnancy test in urine or blood

Exclusion Criteria:

* Women currently pregnant or in the lactation period.
* Patients whose companion is pregnant.
* Therapy with interferon (IFN) or ribavirin at any previous time.
* Patients with cirrhosis in the hepatic biopsy.
* Documented suspicion by ultrasound of hepatocarcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with undetectable RNA-HCV | at week 12 after starting treatment

SECONDARY OUTCOMES:
Variations of the levels of RNA-HCV | from baseline until weeks 4, 8, and 12 of the study
Percentage of patients with undetectable HCV RNA | in weeks 4 and 8 of the study
Levels of ALT | At weeks 4, 8, and 12
Percentage of patients that must reduce the dose of peginterferon alpha-2a (40 KD) and ribavirin. | During the 12 weeks of follow-up
Percentage of patients that drop out of the study for adverse effects or intolerance | During the 12 weeks of follow-up
Variations in levels of haemoglobin, neutrophil, and platelet count | at 4, 8, and 12 weeks with regard to baseline
AIDS-defining events or death | During the 12 weeks of follow-up
Changes in the CD4/CD8 cell count | At 4, 8, and 12 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit
Locations (12):
- Spain (12):
  - Hospital Germans Trias i Pujol, Badalona, Badalona, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital General de Vic, Vic, Barcelona
  - Hospital de Donostia, San Sebastián, Donostia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Gregorio Marañón., Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid